CLINICAL TRIAL: NCT00061672
Title: A Phase II Study Evaluating the Safety and Effectiveness of ABT-510 in Subjects With Refractory Lymphoma
Brief Title: Study Evaluating the Safety and Effectiveness of ABT-510 in Subjects With Refractory Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-457
Record Dates: First submitted 2003-06-02; First posted 2003-06-04 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma (NHL); Hodgkin's Lymphoma (HL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-510 - Thrombospondin-1 Mimetic

SUMMARY:
The primary objective of this study is to assess the safety and effectiveness of ABT-510 in subjects with refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if all of the following criteria are met:

* The subject is at least 18 years of age.
* The subject has histologically confirmed non-Hodgkin's Lymphoma (NHL) (excluding Burkitt's, Burkitt's type or HIV associated lymphoma) or Hodgkin's Lymphoma (HL) that is refractory to or has relapsed after standard therapy or for which there is no known effective treatment.
* The subject must have measurable disease by the CHESON Criteria for Tumor Response.
* The subject has an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
* The subject is able to self-administer or has a caregiver who can reliably administer subcutaneous injections.
* The subject must have adequate bone marrow, renal and hepatic function as follows:

  * Bone marrow: *White blood cell count (WBC) greater than or equal to 3,000/mm3; *Platelets greater than or equal to 75,000/mm3 unless subject has received a prior transplant or bone marrow involvement with lymphoma has been documented, then platelets of equal to or greater than 50,000 is acceptable. *Hemoglobin greater than or equal to 8.5 g/dL; *ANC greater than or equal to 1000/mm3
  * Renal function: *Serum creatinine less than or equal to 2.0 mg/dL
  * Hepatic function: *AST and ALT less than or equal to 3.0 X ULN
* The subject must not be pregnant or lactating and all subjects (male and female) must use a contraceptive method deemed appropriate by the investigator while in the study and up to two months following completion of therapy.
* The subject has voluntarily signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved consent prior to any study specific procedures.

Exclusion Criteria:

A subject will be ineligible for study participation if any of the following criteria are met:

* The subject has a history of or currently exhibits Central Nervous System (CNS) metastasis. Brain MRI within 28 days of enrollment is required to confirm absence of CNS metastases.
* The subject is receiving therapeutic anticoagulation therapy. Low dose anticoagulation (e.g., low dose Coumadin) for catheter prophylaxis is permitted; PT/PTT must be within normal limits.
* The subject has a history of or currently exhibits clinically significant cancer related events of bleeding (e.g., hemoptysis). The subject has a recent history of (within 4 weeks of Study Day 1) or currently exhibits other clinically significant events of bleeding.
* The subject has received any therapy for lymphoma including chemotherapy, antibody therapy, radiotherapy or any investigational therapy within four weeks prior to study drug administration.
* The subject has been initiated on steroids or there is an increase in current steroid dose within three months prior to study drug administration.
* The subject exhibits evidence of clinically significant uncontrolled condition(s) and/or is considered by the investigator to be unable to tolerate the proposed treatment or procedures.
* The subject has history of other previous malignancies within 5 years, with the exception of: Adequately treated in situ carcinoma of the cervix; Basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2003-04

PRIMARY OUTCOMES:
Response rate | One year

SECONDARY OUTCOMES:
Progression free survival | One year
Overall survival | One year
Performance status | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rod Humerickhouse, MD, Study Director — Abbott
Locations (14):
- United States (14):
  - Hematology Oncology Associates, Phoenix, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - USC - Norris Cancer Center, Los Angeles, California
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Cancer Centers of Florida, P.A., Orlando, Florida
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Arch Medical Services, INC., St Louis, Missouri
  - Albany Regional Cancer Center, Albany, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - The West Cancer Clinic, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Hematology Oncology Associates, San Antonio, Texas
  - U of W - Comprehensive Care Center, Madison, Wisconsin